CLINICAL TRIAL: NCT07069543
Title: Changes in Polysomnography and Rhinomanometry Parameters After Rapid Maxillary Expansion or Adenotonsilectomy in Children With Sleep Apnea
Brief Title: Changes in Polysomnography and Rhinomanometry Parameters After Rapid Maxillary Expansion or Adenotonsilectomy in Children With Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Mariana Maciel Tinano, Associate Professor, Outpatient clinic for the Mouth-breathers,, Federal University of Minas Gerais
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: COEP/UFMG number 51038721.7.00
Record Dates: First submitted 2025-06-02; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Obstructive Sleep Apnea (OSA); Rapid Maxillary Expansion; Polysomnography
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: A sample of 51 children aged 5 to 10 years, diagnosed with OSA through PSG and referred for AT, was selected in a hospital based mouth-breathing specialized center. Children were divided in 2 groups: the AT group with 25 individuals, without maxillary hypoplasia, and the RME group composed of 26 children with maxillary constriction and posterior crossbite, with indication for RME before the AT surgery. Children underwent an initial evaluation at the time of selection (T0) and six months after the intervention: AT or RME (T1).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adenotonsillectomy group (Experimental): adenotonsillectomy surgical group
  Interventions: Procedure: Adenotonsillectomy
- Rapid maxillary expansion group (Experimental): rapid maxillary expansion group
  Interventions: Procedure: Rapid maxillary expansion

INTERVENTIONS:
Procedure: Adenotonsillectomy — the adenotonsillectomy group children, indicated for immediate adenotonsillectomy
  Arms: Adenotonsillectomy group
Procedure: Rapid maxillary expansion — expansion group children with a narrow palate and posterior crossbite, with indication for rapid maxillary expansion
  Arms: Rapid maxillary expansion group

SUMMARY:
Adenotonsillectomy (AT) is considered the most effective and the standard treatment for Obstructive Sleep Apnea (OSA) in children. Since maxillary hypoplasia is a risk factor for OSA, Rapid Maxillary Expansion (RME) has been be considered as a complementary treatment in selected cases,improving the OSA. To compare changes in polysomnography (PSG) and in anterior active rhinomanometry (AAR) in children diagnosed with OSA, treated with RME or AT.

Methods: A sample of 51 children aged 5 to 10 years, diagnosed with OSA through PSG and referred for AT, was selected in a hospital based mouth-breathing specialized center. Children were divided in 2 groups: the AT group with 25 individuals, without maxillary hypoplasia, and the RME group composed of 26 children with maxillary constriction and posterior crossbite, with indication for RME before the AT surgery. Children underwent an initial evaluation at the time of selection (T0) and six months after the intervention: AT or RME (T1).

DETAILED DESCRIPTION:
PSG was performed to measure the apnea/hypopnea index (AHI), mean and minimum oxygen saturation (SpO2), desaturation index and desaturation time below 90%. AAR was used to measure nasal inspiratory flow (NIF), % NIF and nasal resistance. To compare the differences between the groups at T0, T1 and T1-T0, t-tests and Mann-Whitney tests were used. To compare the changes resulting from ERM and AT, paired t-tests and the Wilcoxon test were used, for a statistical significance level of 5%.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of OSA confirmed by polysomnography
* between 5 and 10 years of age
* Indication for adenotonsillectomy (adenoids occupying more than 75% of the nasopharynx and/or tonsils classified as degree 3 or 4)

Exclusion Criteria:

* Children with systemic diseases
* craniofacial syndromes that interfered with functional and psychosocial development,
* children who did not complete the expansion
* parents did not sign the informed consent

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2024-03-02 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
polysomnography measures | Children underwent at enrollment (T0) and six months after the intervention: AT or RME (T1).
  PSG was performed to measure the apnea/hypopnea index (AHI)
polysomnography measures | Children underwent at enrollment (T0) and six months after the intervention: AT or RME (T1).
  PSG was performed to measure the mean and minimum oxygen saturation (SpO2)
polysomnography measures | Children underwent at enrollment (T0) and six months after the intervention: AT or RME (T1).
  PSG was performed to measure the desaturation index
polysomnography measures | Children underwent at enrollment (T0) and six months after the intervention: AT or RME (T1).
  PSG was performed to measure the desaturation time below 90%.

SECONDARY OUTCOMES:
anterior active rhinomanometry measures | Children underwent at enrollment (T0) and six months after the intervention: AT or RME (T1).
  AAR was used to measure the nasal inspiratory flow (NIF)
anterior active rhinomanometry measures | Children underwent at enrollment (T0) and six months after the intervention: AT or RME (T1).
  AAR was used to measure the nasal inspiratory flow percent (NIF)
anterior active rhinomanometry measures | Children underwent at enrollment (T0) and six months after the intervention: AT or RME (T1).
  AAR was used to measure the nasal resistance.

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Minas Gerais, Belo Horizonte, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: Yes
only IPD used in the results publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years after the publication of results
Access Criteria: Statistical analyses of the study results will be shared through Excel spreadsheets